CLINICAL TRIAL: NCT02083380
Title: Randomised Phase IIb Study of Efficacy, Safety, Tolerability & Pharmacokinetics of a Single Dose Regimen of Artefenomel (OZ439) in Loose Combination With Piperaquine in Adults and Children With Uncomplicated Plasmodium Falciparum Malaria.
Brief Title: Phase II Efficacy Study of Artefenomel & Piperaquine in Adults & Children With P. Falciparum Malaria.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV_OZ439_13_003
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: Plasmodium falciparum malaria; malaria; OZ439; piperaquine; PQP
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — artefenomel; piperaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A) Artefenomel 800mg: piperaquine 640mg (Experimental): One single dose of Artefenomel 800mg: Piperaquine phosphate 640mg loose combination
  Interventions: Drug: Artefenomel 800mg: piperaquine 640mg
- B) Artefenomel 800mg: piperaquine 960mg (Experimental): One single dose of Artefenomel 800mg: Piperaquine phosphate 960mg loose combination
  Interventions: Drug: Artefenomel 800mg: piperaquine 960mg
- C) Artefenomel 800mg: piperaquine 1440mg (Experimental): One single dose of Artefenomel 800mg: Piperaquine phosphate 1440mg loose combination
  Interventions: Drug: Artefenomel 800mg: piperaquine 1440mg

INTERVENTIONS:
Drug: Artefenomel 800mg: piperaquine 640mg — Active, loose combination
  Other Names: OZ439 ; PQP
  Arms: A) Artefenomel 800mg: piperaquine 640mg
Drug: Artefenomel 800mg: piperaquine 960mg — Active, loose combination
  Other Names: OZ439 ; PQP
  Arms: B) Artefenomel 800mg: piperaquine 960mg
Drug: Artefenomel 800mg: piperaquine 1440mg — Active, loose combination
  Other Names: OZ439 ; PQP
  Arms: C) Artefenomel 800mg: piperaquine 1440mg

SUMMARY:
A randomised, double-blind single-dose study to determine the efficacy, safety, tolerability and pharmacokinetics of OZ439 (artefenomel) in combination with piperaquine (PQP) in patients > 0.5 years and <= 70 years of age with uncomplicated Plasmodium falciparum malaria in Africa and Asia (Vietnam).

Interim analyses for futility were planned. Adults and children will be included through progressive step-down in age following safety review by an independent safety monitoring board (ISMB).

If the study were to meets its efficacy objectives, this will inform dose setting for Phase III studies.

DETAILED DESCRIPTION:
A randomised, double-blind single-dose (loose combination) study in the target patient population of children > 0.5 years and <= 5 years of age in Africa and patients of all ages in Asia (> 0.5 years and <= 70 years) with uncomplicated Plasmodium falciparum malaria. Patients > 5 years in Africa were also to be recruited in a safety age step down procedure. The underlying assumption was that children of 5 years or less in Africa and all ages in Asia will have a higher probability of having lower immunity and hence potentially require higher drug exposure to achieve efficacy and hence the study aimed to recruit 60-80% African children < = 5 years and 18-36% Asian patients (defined as the target population) and approximately 10% African patients >5 years,

Three OZ439/PQP treatment arms were to be included for patients >= 35 kg (800mg OZ439 in loose combination with PQP doses of either 640, 960, 1440 mg). Doses were scaled for patients < 35kg based on the weight to achieve similar exposures in patients >= 35kg.

The study was to test for futility and dose arms were to be dropped if the probability was >30% that PCR-adjusted ACPR at Day 28 (ACPR28) was less than 90% (the target efficacy for the study was >= 95% ACPR28). Only data from patients in Asia patients and Africa patients < 5 years were to be included in the Interim analysis, although all patients were to be included in the final analysis. Interim analyses were to occur after recruitment of approximately 50 evaluable patients per dose cohort and thereafter approximately after every 25 patients.

In a separate process, the safety of OZ439/PQP treatment arms was to be assessed at scheduled time points by an ISMB and adults and children were included through progressive step-down in age range following safety evaluation

Following Screening and informed consent, patients were to receive study drug and were to be followed for clinical signs of malaria (parasitaemia and temperature), safety assessments and pharmacokinetics up to Day 42 following dosing (Day 63 at selected sites).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient age >6 months <70 years.
2. Body weight >5 kg <90 kg.
3. Presence of mono-infection of P. falciparum with:

   1. Fever, as defined by axillary temperature ≥ 37.5°C or oral/rectal/tympanic temperature ≥ 38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
   2. Microscopically confirmed parasite infection, in range 1,000 to 100,000 asexual parasites /µL of blood.
4. Written informed consent provided by the adult patient, or parent or legally acceptable representative (LAR) of the minor patient or by an impartial witness (if the patient or patient's LAR is illiterate), and by the medically qualified Investigator. Children will be asked to provide assent where appropriate. The age from which this will be sought will be defined by local legislation.

Exclusion Criteria:

1. Presence of severe malaria (according to World Health Organization (WHO) definition - WHO 2013)
2. Anti-malarial treatment:

   1. With piperaquine -based compound, mefloquine, naphthoquine or sulphadoxine/pyrimethamine (SP) within the previous 6 weeks (after their inhibition of new infections has fallen below 50%).
   2. With amodiaquine or chloroquine within the previous 4 weeks.
   3. With quinine, halofantrine, lumefantrine-based compounds and any other anti-malarial treatment or antibiotics with anti-malarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones, and azithromycin) within the past 14 days.
   4. With any herbal products or traditional medicines, within the past 7 days.
3. Known history or evidence of clinically significant disorders such as, respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological, neurological (including auditory), endocrine, infectious, malignancy, psychiatric, history of convulsions or other abnormality (including head trauma).
4. Family history of sudden death or of congenital or clinical conditions known to prolong QTcB or QTcF interval or e.g. patients with a history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease.
5. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
6. Any predisposing cardiac conditions for arrhythmia such as severe hypertension, left ventricular hypertrophy (including hypertrophic cardiomyopathy) or congestive cardiac failure accompanied by reduced left ventricle ejection fraction.
7. Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia or hypomagnesaemia.
8. Any treatment which can induce a lengthening of QT interval, such as:

   1. Antiarrhythmics (e.g. amiodarone, disopyramide, dofetilide, ibutilide, procainamide, quinidine, hydroquinidine, sotalol),
   2. Neuroleptics (e.g. phenothiazines, sertindole, sultopride, chlorpromazine, haloperidol, mesoridazine, pimozide, or thioridazine),
   3. Anti-depressive agents, certain antimicrobial agents, including agents of the following classes macrolides (e.g. erythromycin, clarithromycin), fluoroquinolones (e.g. moxifloxacin, sparfloxacin), imidazole and triazole antifungal agents, and also pentamidine and saquinavir,
   4. Certain non-sedating antihistamines (e.g. terfenadine, astemizole, mizolastine), cisapride, droperidol, domperidone, bepridil, diphemanil, probucol, levomethadyl, methadone, vinca alkaloids, arsenic trioxide.
   5. Anti-emetics with known QT prolongation potential such as domperidone
9. Mixed Plasmodium infection
10. Severe vomiting, defined as more than three times in the 24 hours prior to enrolment in the study or inability to tolerate oral treatment, or severe diarrhoea defined as 3 or more watery stools per day
11. Severe malnutrition (defined for subjects aged ten years or less as the weight-for-height being below -3 standard deviation or less than 70% of median of the National Centre for Health Statistics (NCHS)/WHO normalised reference values, and for subjects aged greater than ten years, a body mass index (BMI) of less than 16 (WFP Manual, Chapter 1)).
12. Known history of hypersensitivity, allergic or adverse reactions to piperaquine or other aminoquinolones or to OZ439 or OZ277
13. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab).
14. If Total Bilirubin is normal, exclude the patient if liver function tests Aspartate transaminase (AST)/ Alanine transaminase (ALT) ≥ 2x Upper limit of normal (ULN).
15. If Total Bilirubin is > 1 and ≤ 1.5xULN, exclude the patient if AST/ALT >1.5xULN.
16. Total Bilirubin > 1.5XULN
17. Haemoglobin level below 8 g/dL.
18. Serum creatinine levels ≥2 x ULN
19. Female patients of child bearing potential must be neither pregnant (as demonstrated by a negative pregnancy test) nor lactating, and must be willing to take measures not to become pregnant during the study period and safety follow-up period.
20. Have received an investigational drug within the past 4 weeks.
21. Previous participation in any malaria vaccine study or received malaria vaccine in any other circumstance.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Macintyre, PhD, Study Director — Medicines for Malaria Venture; Michael Ramharter, MD, Principal Investigator — CERMEL (Centre de Recherches Médicale de Lambaréné)
Locations (9):
- Centre D'Étude Et de Recherchesur Le Paludisme Associé À La Grossesse Et À L'Enfance (Cerpage) Cerpage, Cotonou, Benin
- Burkina Faso (2):
  - Centre National de Recherche et de Formation sur le paludisme (CNRFP) Ouagadougou, Kadiogo, Ouagadougou
  - Clinical research Unit of Nanoro (CRUN)/CMA Saint Camille de Nanoro, 11 BP 218 Ouagadougou CMS 11, Ouagadougou
- Kinshasa School of Public Health, School of Medicine University of Kinshasa, Kinshasa, Democratic Republic of the Congo
- Gabon (2):
  - Centre de Recherches Medicales de Lambarene, Albert Schweitzer Hospital, Lambaréné
  - arielle K. Bouyou-Akotet, Department of Parasitology-Mycology and Tropical Medicine, Faculty of Medicine, Université des Sciences de la Santé, BP 4009, Libreville, Gabon, Libreville
- MANHIÇA HEALTH RESEARCH CENTER, Rua 12, Vila da Manhica, Maputa,, Chefe Maputa, Mozambique
- Tororo District Hospital, Tororo, Uganda
- National Institute of Malariology, Parasitology and Entomology, 245 Luong The Vinh Street, Trung van, Tu Liem, Hanoi, Vietnam, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leroy D, Macintyre F, Adoke Y, Ouoba S, Barry A, Mombo-Ngoma G, Ndong Ngomo JM, Varo R, Dossou Y, Tshefu AK, Duong TT, Phuc BQ, Laurijssens B, Klopper R, Khim N, Legrand E, Menard D. African isolates show a high proportion of multiple copies of the Plasmodium falciparum plasmepsin-2 gene, a piperaquine resistance marker. Malar J. 2019 Apr 10;18(1):126. doi: 10.1186/s12936-019-2756-4. PMID 30967148
- [Derived] Macintyre F, Adoke Y, Tiono AB, Duong TT, Mombo-Ngoma G, Bouyou-Akotet M, Tinto H, Bassat Q, Issifou S, Adamy M, Demarest H, Duparc S, Leroy D, Laurijssens BE, Biguenet S, Kibuuka A, Tshefu AK, Smith M, Foster C, Leipoldt I, Kremsner PG, Phuc BQ, Ouedraogo A, Ramharter M; OZ-Piperaquine Study Group. A randomised, double-blind clinical phase II trial of the efficacy, safety, tolerability and pharmacokinetics of a single dose combination treatment with artefenomel and piperaquine in adults and children with uncomplicated Plasmodium falciparum malaria. BMC Med. 2017 Oct 9;15(1):181. doi: 10.1186/s12916-017-0940-3. PMID 28988541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized double blind study. Conduct was July 2014-August 2015 in Africa (Benin, Burkina Faso, Democratic Republic of Congo, Gabon, Mozambique and Uganda) and Vietnam. Following informed consent patients were recruited to the study. Patients below the age to give legal Informed Consent were consented according local customs / legal requirements.
Pre-assignment Details: Patients were assigned a screening number and underwent screening procedures to assess eligibility. Eligible patients were randomized through an Interactive web-response system and followed for efficacy and safety up to 42 days post dose and 63 days at selected centers. Patients were consented separately to remain in the study up to Day 63.
Groups:
- A) Artefenomel 800mg: Piperaquine 640mg: Artefenomel 800mg: Piperaquine phosphate 640mg loose combination
- B) Artefenomel 800mg: Piperaquine 960mg: Artefenomel 800mg: Piperaquine phosphate 960mg loose combination
- C) Artefenomel 800mg: Piperaquine 1440mg: Artefenomel 800mg: Piperaquine phosphate 1440mg loose combination
Period: Overall Study
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Started | 148 (5 subjects excluded from safety / ITT population - no drug administered) | 151 (3 subjects excluded from safety / ITT population - no drug administered) | 149 (3 subjects excluded from safety / ITT population - no drug administered)
Completed (Lack of Efficacy = Received rescue treatment therefore linked with the efficacy endpoint ACPR) | 57 | 56 | 65
Not Completed | 91 | 95 | 84
Not completed — Lack of Efficacy | 68 | 79 | 64
Not completed — Withdrawal by Subject | 9 | 3 | 7
Not completed — Physician Decision | 1 | 6 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 5 | 3 | 3
Not completed — Other | 8 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- A) Artefenomel 800mg: PQP 640mg: Artefenomel 800mg: Piperaquine 640mg
- B) Artefenomel 800mg: PQP 960mg: Artefenomel 800mg: Piperaquine 960mg
- C) Artefenomel 800mg: PQP 1440mg: Artefenomel 800mg: Piperaquine 1440mg
- Total: Total of all reporting groups
Arm/Group | A) Artefenomel 800mg: PQP 640mg | B) Artefenomel 800mg: PQP 960mg | C) Artefenomel 800mg: PQP 1440mg | Total
Number analyzed (Participants) | 143 | 148 | 146 | 437
Age, Customized [Number; unit: participants]
  > 15 years | 41 | 42 | 41 | 124
  > 5 to <= 15 years | 8 | 8 | 9 | 25
  > 2 to <= 5 years | 69 | 72 | 70 | 211
  >= 0.5 to <= 2 years | 25 | 26 | 26 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 98 | 266
  Male | 60 | 63 | 48 | 171

OUTCOME MEASURES:

1. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population (All Patients)
Description: Polymerase chain reaction (PCR)-adjusted adequate clinical and parasitological response (ACPR) at Day 28: defined as: absence of parasitaemia on Day 28, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure (ETF), late clinical failure (LCF) or late parasitological failure (LPF). Definition of ETF, LCF and LPF according to a modified standard WHO classification. Per protocol population (PP).
  95% Clopper-Pearson 2-sided Confidence Interval (CI) constructed around the single binomial proportion per treatment arm and total.
Time Frame: Day 28
Population: Primary analysis population was the per protocol population defined as all patients comprising the ITT set and without major protocol deviations. Including insufficient evidence of study indication, no baseline parasitemia and non-compliance with study drug administration.
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 106 | 117 | 117
% ACPR PCR-adjusted | 70.8 [61.13 to 79.19] | 68.4 [59.13 to 76.66] | 78.6 [70.09 to 85.67]

2. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population: Asia (All Ages)
Description: PCR-adjusted adequate clinical and parasitological response (ACPR) at Day 28: defined as: absence of parasitaemia on Day 28, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure (ETF), late clinical failure (LCF) or late parasitological failure (LPF). Definition of ETF, LCF and LPF according to a modified standard WHO classification.
  95% Clopper-Pearson 2-sided CI constructed around the single binomial proportion per treatment arm and total.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 25 | 25 | 27
% ACPR PCR-adjusted | 64 [42.52 to 82.03] | 64 [42.52 to 82.03] | 70.4 [49.82 to 86.25]

3. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population: Africa (All Ages)
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 81 | 92 | 90
% ACPR PCR-adjusted | 72.8 [61.81 to 82.13] | 69.6 [59.10 to 78.73] | 81.1 [71.49 to 88.59]

4. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population: Africa (> Than 5 Years)
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 18 | 21 | 19
% ACPR PCR-adjusted | 77.8 [52.36 to 93.59] | 90.5 [69.62 to 98.83] | 89.5 [66.86 to 98.70]

5. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population: Africa (< = 5 Years)
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 63 | 71 | 71
% ACPR PCR-adjusted | 71.4 [58.65 to 82.11] | 63.4 [51.10 to 74.50] | 78.9 [67.56 to 87.67]

6. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population: Africa (>2 to <= 5 Years)
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 45 | 50 | 55
% ACPR PCR-adjusted | 75.6 [60.46 to 87.12] | 74.0 [59.66 to 85.37] | 83.6 [71.20 to 92.23]

7. Primary Outcome: PCR-adjusted ACPR at Day 28 in the PP Population: Africa (>= 0.5 to <= 2 Years)
Description: as for outcome 2
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 18 | 21 | 16
% ACPR PCR-adjusted | 61.1 [35.75 to 82.70] | 38.1 [18.11 to 61.56] | 62.5 [35.43 to 84.80]

8. Secondary Outcome: PCR - Adjusted ACPR at Day 42 in the PP Population
Description: PCR - adjusted adequate clinical and parasitological response at Day 42
Time Frame: Days 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 100 | 108 | 100
% ACPR PCR-adjusted | 65.0 [54.82 to 74.27] | 65.7 [55.99 to 74.60] | 72.0 [62.13 to 80.52]

9. Secondary Outcome: PCR-adjusted ACPR at Day 63 in the PP Population
Description: PCR-adjusted adequate clinical and parasitological response at Day 63
Time Frame: Day 63
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 83 | 90 | 84
% ACPR PCR-adjusted | 57.8 [46.49 to 68.60] | 58.9 [48.02 to 69.16] | 69.0 [58.02 to 78.69]

10. Secondary Outcome: Crude ACPR at Day 28 in the PP Population
Description: Crude adequate clinical and parasitological response at Day 28
Time Frame: Day 28
Population: Primary analysis population was the per protocol population defined as all patients comprising the ITT set and without major protocol deviations. Including insufficient evidence of study indication, no baseline parasitemia and non-compliance with study drug administration. The PP population comprised 93.3% of the randomized population.
Measure: Number (95% Confidence Interval); unit: % ACPR unadjusted (crude)
Groups:
- C) Artefenomel 800mg: Piperaquine 1440mg: C) Artefenomel 800mg: Piperaquine phosphate 1440mg loose combination
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 129 | 136 | 133
% ACPR unadjusted (crude) | 57.4 [48.36 to 66.03] | 56.6 [47.85 to 65.09] | 66.9 [58.23 to 74.83]

11. Secondary Outcome: Crude ACPR at Day 42 in the PP Population
Description: Crude adequate clinical and parasitological response at Day 42
Time Frame: Day 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % ACPR unajusted (crude)
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 127 | 134 | 130
% ACPR unajusted (crude) | 48.0 [39.09 to 57.07] | 48.5 [39.79 to 57.29] | 51.5 [42.62 to 60.39]

12. Secondary Outcome: Crude ACPR at Day 63 in the PP Population
Description: Crude adequate clinical and parasitological response at Day 63
Time Frame: Day 63
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: % ACPR unadjusted (crude)
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 114 | 122 | 116
% ACPR unadjusted (crude) | 42.1 [32.92 to 51.71] | 39.3 [30.62 to 48.59] | 49.1 [39.74 to 58.58]

13. Secondary Outcome: PCR-adjusted ACPR at Day 28 in the ITT Population
Description: PCR-adjusted adequate clinical and parasitological response at Day 28. Intent to Treat ( ITT) population.
Time Frame: Day 28
Population: Intent to Treat (ITT) population : all patients who provided written informed consent, were randomised, received the single dose combination of OZ439/PQP study drug (or part thereof), and had a confirmed positive blood film for P. falciparum asexual parasitaemia at inclusion.
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 143 | 148 | 146
% ACPR PCR-adjusted | 53.8 [45.32 to 62.21] | 55.4 [47.02 to 63.57] | 65.1 [56.75 to 72.76]

14. Secondary Outcome: PCR-adjusted ACPR at Day 42 in the ITT Population
Description: PCR-adjusted adequate clinical and parasitological response at Day 42 in the ITT population
Time Frame: Day 42
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 143 | 148 | 146
% ACPR PCR-adjusted | 46.9 [38.47 to 55.37] | 48.6 [40.36 to 56.99] | 50.0 [41.62 to 58.38]

15. Secondary Outcome: PCR-adjusted ACPR at Day 63 in the ITT Population
Description: PCR-adjusted adequate clinical and parasitological response at Day 63 in the ITT population
Time Frame: Day 63
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: % ACPR PCR-adjusted
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 136 | 140 | 135
% ACPR PCR-adjusted | 36.8 [28.67 to 45.45] | 38.6 [30.47 to 47.16] | 43.7 [35.19 to 52.50]

16. Secondary Outcome: Crude ACPR at Day 28 in the ITT Population
Description: Crude adequate clinical and parasitological response at Day 28 in the ITT population
Time Frame: Day 28
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: % ACPR unadjusted (crude)
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 143 | 148 | 146
% ACPR unadjusted (crude) | 53.1 [44.63 to 61.53] | 53.4 [45.01 to 61.61] | 63.0 [54.64 to 70.85]

17. Secondary Outcome: Crude ACPR at Day 42 in the ITT Population
Description: Crude adequate clinical and parasitological response at Day 42 in the ITT population
Time Frame: Day 42
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: % ACPR unadjusted (crude)
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 143 | 148 | 146
% ACPR unadjusted (crude) | 44.1 [35.77 to 52.59] | 44.6 [36.43 to 52.98] | 46.6 [38.29 to 55.01]

18. Secondary Outcome: Crude ACPR at Day 63 in the ITT Population
Description: Crude adequate clinical and parasitological response at Day 63 in the ITT population
Time Frame: Day 63
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: % ACPR unadjusted (crude)
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 136 | 140 | 135
% ACPR unadjusted (crude) | 36.8 [28.67 to 45.45] | 35.0 [27.14 to 43.51] | 43.0 [34.48 to 51.76]

19. Secondary Outcome: Kaplan-Meier Estimate of Recurrence
Description: Kaplan-Meier estimate of number of recurrent infections (either recrudescence or new infection)
Time Frame: Day 63
Population: modified Intent to Treat (mITT) population : all patients who provided written informed consent, were randomised, were compliant with the single dose combination of OZ439/PQP study drug and had a confirmed positive blood film for P. falciparum asexual parasitaemia at inclusion.
Measure: Number; unit: % population recurring
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 141 | 141 | 140
% population recurring | 44.7 | 54.6 | 43.6

20. Secondary Outcome: Kaplan-Meier Estimate of Recrudescence
Description: Kaplan-Meier estimate of number of patients with recrudescence
Time Frame: Day 63
Population: as for outcome 19
Measure: Number; unit: % patients with recrudescence
Groups:
- A) Arttefenomel 800mg: Piperaquine 640mg: Artefenomel 800mg: Piperaquine phosphate 640mg loose combination
Arm/Group | A) Arttefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 141 | 141 | 140
% patients with recrudescence | 22.7 | 29.1 | 18.6

21. Secondary Outcome: Kaplan-Meier Estimate of New Infection Rate
Description: Kaplan-Meier estimate of number of patients with new infections
Time Frame: Day 63
Population: as for outcome 19
Measure: Number; unit: % population with new infection
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 141 | 141 | 140
% population with new infection | 11.3 | 16.3 | 13.6

22. Secondary Outcome: Parasite Clearance Time
Description: Time post dose to parasite clearance
Time Frame: 0, 6, 12, 18, 24, 30, 36, 48 and 72 hours post dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 139 | 140 | 139
hours | 36.1 [36.0 to 36.1] | 36.0 [36.0 to 36.1] | 36.1 [36.0 to 36.1]

23. Secondary Outcome: Fever Clearance Time
Description: Time to fever clearance (hours)
Time Frame: Day 42
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 139 | 140 | 139
hours | 1.0 [1.0 to 2.6] | 1.2 [1.0 to 2.1] | 1.1 [1.0 to 2.0]

24. Secondary Outcome: PRR48
Description: Parasite reduction ratio at 48 hours post dose
Time Frame: 0, 6, 12, 18, 24, 30, 36 and 48 hours post dose
Population: Primary analysis population was the per protocol population defined as all patients comprising the ITT set and without major protocol deviations. Including insufficient evidence of study indication, no baseline parasitemia and non-compliance with study drug administration. Subjects with sufficient data points to determine PRR48
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 97 | 103 | 99
ratio | 9.120 [6.900 to 12.970] | 9.300 [7.660 to 13.340] | 8.690 [6.850 to 12.260]

25. Other Pre Specified Outcome: Piperaquine: Cday7 Asia (All Ages)
Description: Piperaquine concentration at Day7 in Asian patients all ages
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 27 | 28 | 28
ng/mL | 4.2 (72) | 6.9 (61) | 9.3 (78)

26. Other Pre Specified Outcome: Piperaquine: Cday7 Africa (> 5 Years)
Description: Piperaquine concentration at Day7 in African patients > 5 years
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 21 | 22 | 21
ng/mL | 5.6 (113) | 8.8 (105) | 12.1 (103)

27. Other Pre Specified Outcome: Piperaquine: Cday7 Africa (>2 to <= 5 Years)
Description: Piperaquine concentration at Day7 in African patients > 2 and <= 5years
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 43 | 42 | 33
ng/mL | 6.3 (71) | 9.2 (87) | 10.9 (92)

28. Other Pre Specified Outcome: Piperaquine: Cday7 Africa (>=0.5 to <= 2 Years)
Description: Piperaquine concentration at Day7 in African patients >= 0.5 and <= 2 years
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A) Artefenomel 800mg: Piperaquine 640mg | B) Artefenomel 800mg: Piperaquine 960mg | C) Artefenomel 800mg: Piperaquine 1440mg
Number analyzed (Participants) | 51 | 52 | 59
ng/mL | 5.0 (63) | 5.9 (70) | 9.0 (94)

29. Other Pre Specified Outcome: Artefenomel Cday7 Asian Patients (All Ages)
Description: Artefenomel concentration on Day 7 in Asian Patients (all ages). All Treatment arms.
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- A) Artefenomel 800mg: PQP 640mg, 960mg & 1440mg: Artefenomel 800mg: Piperaquine phosphate 640mg, 960mg & 1440mg combined
  Artefenomel 800mg: PQP 640mg, 960mg & 1440mg
Arm/Group | A) Artefenomel 800mg: PQP 640mg, 960mg & 1440mg
Number analyzed (Participants) | 82
ng/mL | 5.1 (95)

30. Other Pre Specified Outcome: Artefenomel Cday7 African Patients (> 5 Years)
Description: Artefenomel concentration on Day 7 in African Patients > 5 years. All Treatment arms.
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- A) Artefenomel 800mg: PQP 640mg, 960mg & 1440mg: Artefenomel 800mg: Piperaquine phosphate 640mg, 960mg & 1440mg combined
Arm/Group | A) Artefenomel 800mg: PQP 640mg, 960mg & 1440mg
Number analyzed (Participants) | 64
ng/mL | 3.3 (141)

31. Other Pre Specified Outcome: Artefenomel Cday7 African Patients (>2 to <= 5 Years)
Description: Artefenomel concentration on Day 7 in African Patients >2 to <= 5 years. All Treatment arms.
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A) Artefenomel 800mg: PQP 640mg, 960mg & 1440mg
Number analyzed (Participants) | 120
ng/mL | 3.3 (142)

32. Other Pre Specified Outcome: Artefenomel Cday7 African Patients (>=0.5 to <= 2 Years)
Description: Artefenomel concentration on Day 7 in African Patients >= 0.5 to <=2 years. All Treatment arms.
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A) Artefenomel 800mg: PQP 640mg, 960mg & 1440mg
Number analyzed (Participants) | 161
ng/mL | 2.0 (147)

ADVERSE EVENTS:
Time Frame: From screening up to Day 63 post dose
Groups:
- A) Artefenomel 800mg: PQP 640mg: Artefenomel 800mg: Piperaquine phosphate 640mg
Arm/Group | A) Artefenomel 800mg: PQP 640mg | B) Artefenomel 800mg: PQP 960mg | C) Artefenomel 800mg: PQP 1440mg
Serious Adverse Events (participants affected / at risk) | 1/146 | 1/148 | 2/143
Other Adverse Events (participants affected / at risk) | 122/146 | 127/148 | 115/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A) Artefenomel 800mg: PQP 640mg (N=146) | B) Artefenomel 800mg: PQP 960mg (N=148) | C) Artefenomel 800mg: PQP 1440mg (N=143)
Transaminase elevation (Investigations) | 0 (0) | 0 (0) | 1 (2) — Two reversible SAEs of possibly related reversible transaminase elevation in one subject
Anemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin drop < 5 g/dL (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A) Artefenomel 800mg: PQP 640mg (N=146) | B) Artefenomel 800mg: PQP 960mg (N=148) | C) Artefenomel 800mg: PQP 1440mg (N=143)
malaria (Infections and infestations) | 34 (34) | 45 (48) | 43 (44)
Bronchitis (Infections and infestations) | 10 (11) | 13 (19) | 13 (16)
Rhinitis (Infections and infestations) | 10 (10) | 9 (10) | 11 (11)
Plasmodium Falciparum Infection (Infections and infestations) | 7 (7) | 10 (10) | 9 (9)
Electrocardiumgram QT prolonged (Investigations) | 44 (56) | 41 (48) | 27 (29)
Neutrophil count decreased (Investigations) | 12 (13) | 11 (11) | 18 (18)
Haemoglobin decreased (Investigations) | 11 (11) | 20 (22) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 20 (20) | 21 (21) | 11 (12)
Vomiting (Gastrointestinal disorders) | 16 (16) | 20 (20) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 8 (9) | 5 (5)
Pyrexia (General disorders) | 9 (11) | 12 (13) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No